CLINICAL TRIAL: NCT05712044
Title: Evaluation of the Effect of Folic Acid Supplementation on the Presentation of Nuclear Abnormalities Associated With Cytogenotoxic Damage Induced by Chronic Drug Use.
Brief Title: Effect of Folic Acid on the Presentation of Nuclear Abnormalities in People With a History Drug Abuse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Universitario de Tonalá (Other)
Responsible Party: Principal Investigator, MARIA GUADALUPE SANCHEZ PARADA, Associate professor, Centro Universitario de Tonalá
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F-2022-004
Record Dates: First submitted 2023-01-02; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Drug Abuse; Genotoxicity
MeSH Terms: conditions — Substance-Related Disorders | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study, pretest-posttest design with no control group. equivalent, in subjects with substance abuse and healthy subjects. The intervention will consist of administration of 15 mg of folic acid divided into 3 doses per day. Mucosal samples will be taken orally in duplicate to each participant to determine the frequency of micronuclei (MN), bursts cells (NBUD), binucleated cells (BN), condensed chromatin (CC), karyorrhexis (CR), pyknosis (PIC) and caryolysis (CL) at different time events: pre-treatment, 15 days and 30 days. So as a survey to determine consumption patterns of psychoactives, sociodemographic data, dietary and exposure to known cytogenotoxic agents.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Basal (No Intervention): Samples will be taken to participants.
- 15 days folate suplementation (Experimental): 5mg tablets of folic acid will be given to participants every 8 hours for a period of 15 days, then samples are to be taken in duplicate for each individual.
  Interventions: Drug: Folic Acid 5 MG
- 30 days folate suplementatio (Experimental): 5mg tablets of folic acid will be given to participants every 8 hours fora a period of 30 days, then samples are to be taken in duplicate for each individual.
  Interventions: Drug: Folic Acid 5 MG

INTERVENTIONS:
Drug: Folic Acid 5 MG — Folic acid 5mg tablets will be administered orally every 8 hours then samples from buccal mucosa will be taken 15 days and 30 days after suplementation.
  Other Names: folic acid 5mg cilocid bruluagsa
  Arms: 15 days folate suplementation; 30 days folate suplementatio

SUMMARY:
Background: Multiple studies have pointed to the harmful potential of licit and illicit drugs.

as agents associated with neoplastic processes and other non-communicable diseases, for which reason It has become a problem of global size. Objective: The central objective is to determine the cytogenotoxic damage in the oral mucosa of people with chronic drug use, as well as establishing the therapeutic effect of acid administration folic on said damage. Methodology: Quasi-experimental study, pretest-posttest design with no control group.

equivalent, in subjects with substance abuse and healthy subjects. The intervention will consist of administration of 15 mg of folic acid divided into 3 doses per day. Mucosal samples will be taken orally in duplicate to each participant to determine the frequency of micronuclei (MN), bursts cells (NBUD), binucleated cells (BN), condensed chromatin (CC), karyorrhexis (CR), pyknosis (PIC) and caryolysis (CL) at different time events: pre-treatment, 15 days and 30 days. So as a survey to determine consumption patterns of psychoactives, sociodemographic data, dietary and exposure to known cytogenotoxic agents. Resources and infrastructure: The study will be carried out in the pharmacology laboratory of the Center University of Tonalá, who will make their equipment and reagents available. Group experience: The research group has over a decade of experience in the development of projects related to mutagenesis and cyto-genotoxic agents.

Development time: The project will be developed from February 2023 to August of 2023

DETAILED DESCRIPTION:
Objectives.

* General Objective. To determine the effect of folic acid supplementation on the presentation of nuclear abnormalities associated with cytogenotoxic damage in healthy subjects and chronic drug users.
* Specific objectives.

  1. Determine the presence of micronuclei and other nuclear abnormalities in baseline samples from the group of chronic drug users and the healthy reference group.
  2. To compare baseline cytogenotoxic damage determinations with subsequent damage determinations, at 15 and 30 days, in chronic drug users supplemented with folic acid.

     Material and methods.
* Study design. Quasi-experimental study of pretest-posttest design with non-equivalent control group in subjects with substance abuse and healthy subjects. The intervention will consist of the administration of 15 mg of folic acid divided into 3 doses per day. Duplicate oral mucosa samples will be taken from each participant to determine the frequency of micronuclei (MN), nuclear sprouting (NBUD), binucleated cells (BN), condensed chromatin (CC), karyorrhexis (CR), pyknosis (PIC) and karyolysis. (CL) in different temporary events: pre-treatment, at 15 days and 30 days.

This project will be carried out in inmates of a rehabilitation center in El Salto, Jalisco, Mexico, in participants over 18 years of age, chronic drug users (More than 6 months of consumption). The foregoing under prior informed consent, in a convenience sample of 45 chronic drug users, as well as an equivalent sample of 45 healthy individuals without such a history.

* Sample size At convenience. 45 chronic drug users, inmates of a rehabilitation center in Salto, Jalisco, as well as 45 healthy individuals with no history of drug use will be considered.
* Data collection techniques and instruments. It will be done by taking oral cytology, as well as by means of a confidential questionnaire, in the questionnaire sociodemographic data will be collected such as: sex, age, profession, schooling, as well as information related to the consumption of psychoactive substances such as: tobacco, marijuana, alcohol, inhalants, cocaine and methamphetamines, significant pathological and non-pathological personal history. In addition to data referring to the consumption of a nutritional supplement or vitamin such as folates, B12, C, E, A, lutein or melatonin, or some other antioxidant, medications for pharmacological treatment of chronic disease and/or severe active periodontal disease. Exposure to fertilizers, radiation, heavy metals, as well as place of residence to rule out that they live in areas with high levels of air pollution (Tlaquepaque, Miravalle, Las Juntas and Las Pintas). Likewise, a physical examination of the oral cavity will be carried out by a dentist. All of the above in order to identify pathologies that have been shown to generate bias in the results obtained.

Folic acid will be used in the intervention stage in 5 mg tablets, box with 20 tablets, under the trade name Colicid from Bruluagsa.

---Cyto-genotoxic analysis by micronuclei in exfoliated cells of oral mucosa. The cytogenotoxic effect generated by the drugs will be evaluated, as well as the effect conferred to the administration of folic acid on the presentation of nuclear abnormalities associated with cytogenotoxic damage in chronic drug users.

In supplemented and non-supplemented individuals, through the oral mucosa cell micronucleus bioassay, duplicate samples will be obtained from each individual, spread on slides and stained with specific staining of nucleic acids (NA), frequency of micronuclei (MN), nuclear buds (NBUD), binucleated cells (BN), condensed chromatin (CC), karyorrhexis (CR), pyknosis (PIC) and karyolysis (CL).

---Data management and analysis The analysis of the data will be carried out in the GraphPad 9.2.0 program for Windows. For the continuous quantitative variables, the data will be presented with measures of central tendency and dispersion: mean and standard deviation. For the ordinal quantitative variables, they will be presented in frequencies and percentages, for the comparison of frequencies between sexes and age groups with the Fisher X2 test considering a p < 0.05.

The statistical analysis to find differences between the groups will be carried out by means of the T test and for the ordinal variables it will be calculated by means of Chi2.

ELIGIBILITY:
Inclusion criteria:

* Being 18 years of age or older
* Having used legal and illegal drugs.
* Men or women without diseases

Exclusion criteria:

* People who at the moment of the study or 3 months before:
* Have consumed any dietary supplement or vitamin such as folates, B12,
* C, E, A, lutein or melatonin, or some other antioxidant, medications for
* pharmacological treatment of chronic disease and/or periodontal disease
* severe active.
* That they were exposed to fertilizers, radiation, metals heavy or who live in areas with high levels of air pollution (Tlaquepaque, Miravalle, Las Juntas and Las Pintas).
* Individuals who after have been informed of the advantages and risks of participating in the study, decide not to be part of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Micronucleated cells in 2000 cells | 1 month
  Frequency of micronucleated cells will be assessed in oral mucosa smears for every 2000 cells under fluorescent microscopy, a micronucleated cell has a main nucleus and a smaller one no larger than a third the size of the main nucleus.
Binucleated cells | 1 month
  Frequency of binucleated cells will be assessed in oral mucosa smears for every 2000 cells under fluorescent microscopy, a binucleated cell has two nuclei.
Karyorrhexis | 1 month
  Frequency of karyorrhexis cells will be assessed in oral mucosa smears for every 2000 cells under fluorescent microscopy. Karyorrhexis: cells that appear to have an striated or fragmented nucleus
Karyolysis | 1 month
  Frequency of karyolysis will be assessed in oral mucosa smears for every 2000 cells under fluorescent microscopy. Karyolysis: cells that have lost their nucleus.
Pycnotic nucleus | 1 month
  Frequency of pycnotic cells will be assessed in oral mucosa smears for every 2000 cells under fluorescent microscopy. Pycnotic cells: appear to have a very dense, brighter, and smaller nucleus, approximately one third of the original
Nuclear buds | 1 month
  Frequency of nuclear budding will be assessed in oral mucosa smears for every 2000 cells under fluorescent microscopy. Nuclear bud: a small portion of the genetic material connected through a nucleoplasmic bridge to a main nucleus.
Condensed chromatin | 1 month
  Frequency of condensed chromatin will be assessed in oral mucosa smears for every 2000 cells under fluorescent microscopy. Condensed chromatin: where genetic material can be seen in the nuclei.

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Sanchez, PhD, Principal Investigator — Centro Universitario de Tonalá
Locations (1):
- CUTONALA, Tonalá, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas P, Holland N, Bolognesi C, Kirsch-Volders M, Bonassi S, Zeiger E, Knasmueller S, Fenech M. Buccal micronucleus cytome assay. Nat Protoc. 2009;4(6):825-37. doi: 10.1038/nprot.2009.53. Epub 2009 May 7. PMID 19444240
- [Background] Torres-Bugarin O, Zavala-Cerna MG, Nava A, Flores-Garcia A, Ramos-Ibarra ML. Potential uses, limitations, and basic procedures of micronuclei and nuclear abnormalities in buccal cells. Dis Markers. 2014;2014:956835. doi: 10.1155/2014/956835. Epub 2014 Feb 4. PMID 24778463